CLINICAL TRIAL: NCT02134938
Title: Effects of High-Fibre, Low-Energy Density Viscous Gel Meals on Satiety, Appetite Regulation and Subsequent Food Intake in Healthy Individuals
Brief Title: Effects of Viscous Fibre Containing Foods on Satiety (Gel Form)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: KJM-G
Record Dates: First submitted 2014-04-14; First posted 2014-05-09 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — (1-6)-alpha-glucomannan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Konjac Glucomannan (Experimental): 650g KJM-G
  Interventions: Dietary Supplement: Konjac Glucomannan
- Half Control/Half Konjac Glucomannan (Experimental): 325g KJM-G
  Interventions: Dietary Supplement: Konjac Glucomannan
- Control (No Intervention): 0g KJM-G

INTERVENTIONS:
Dietary Supplement: Konjac Glucomannan — Konjac Noodles (Wellbond Import Export Inc.), Vegan Konjac Shrimp (Sophie's Kitchen), Konjac Gel Cubes
  Arms: Half Control/Half Konjac Glucomannan; Konjac Glucomannan

SUMMARY:
The purpose of this study is to assess whether low caloric, low energy density, konjac food products are effective in appetite regulation when administered as caloric replacements. It is hypothesized that replacement of typical, balanced, vegetarian meals with konjac food products will have comparable satiety scores, decreased postprandial glucose response, and will not significantly affect subsequent food intake.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking males and females
* Aged 18-70 years
* BMI between 18 - 29.9 kg/m²
* Non-dieters (1-10 score on Stunkard Eating Inventory)

Exclusion Criteria:

* Known reported history of liver or kidney disease, diabetes, hypertension, stroke or myocardial infarctions, thyroid disease, Celiac disease/gastrointestinal disease, or AIDS
* Weight change of +/- 3kg in the last 2 months
* Alcohol intake >2 drinks/day
* Inability to consume KJM-G meals
* Any condition which might jeopardize the health and safety of the subject or study personnel, or adversely affect the study results
* Non-compliance with experimental procedures or safety guidelines

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Subjective Satiety | 12 hours for each of the 3 study visits.
  Subjects will record their subjective satiety ratings using a 100 mm visual analogue scale and these ratings will be combined into a total subjective appetite score using the formula (Q1+Q2+(100-Q3)+Q4)/4.

SECONDARY OUTCOMES:
Ambulatory Blood Pressure | Measured at the beginning of each of the 3 study visits and every 30 minutes thereafter until 10:00pm the same day.
Height and Weight | Taken once at the beginning of each of the 3 clinical visits.
Blood Samples | One sample taken immediately prior to (0min) eating each meal (Breakfast, Lunch, Snack and Dinner) and at 30, 60, 90 and 120 min after eating the Breakfast and Lunch meals for each of the 3 study visits (total of 12 blood samples per study visit).
  Capillary blood samples will be collected in anticoagulant containing tubes stored at -20°C and analyzed by trained personnel for plasma glucose concentration using the glucose oxidase method by YSI 2300 STAT Plus within 48 hours.
Palatability Scores | Measured immediately after eating and finishing (<15min after the first bite) each meal (Breakfast, Lunch, Snack and Dinner) for each of the 3 study visits.
Food Craving Rating | Rated immediately prior (0min) to eating each meal (Breakfast, Lunch, Snack and Dinner) for each of the 3 study visits.
  Subjects will record their subjective food craving ratings, if any, prior to each meal, using a 100mm visual analogue scale.
Subsequent Food Intake | Recorded from the 12th to the 24th hour after beginning the first meal (Breakfast at 0min) for each of the 3 study visits.
  Subjects will record their subsequent food intake from 12h to 24h post first meal. Food record will be analyzed with The Nutrition Food Processor (ESHA) and data will be tabulated and included as part of the cumulative daily food intake.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Vuksan, PhD, Principal Investigator — Risk Factor Modification Centre - St. Michael's Hospital; Alexandra Jenkins (Co-Investigator), RD, PhD, Principal Investigator — Risk Factor Modification Centre - St. Michael's Hospital; William Watson (Qualified Investigator), MD, Principal Investigator — Department of Family Medicine - St. Michael's Hospital
Locations (1):
- Clinical Risk Factor and Modification Centre, Toronto, Ontario, Canada